CLINICAL TRIAL: NCT03675139
Title: Medroxyprogesterone Acetate (MPA) Versus Dydrogesterone for Management of Endometrial Hyperplasia Without Atypia
Brief Title: MPA Versus Dydrogesterone for Management of Endometrial Hyperplasia Without Atypia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Principal Investigator, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53201014
Record Dates: First submitted 2018-09-10; First posted 2018-09-18 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Endometrial Hyperplasia Without Atypia
MeSH Terms: interventions — Medroxyprogesterone Acetate; Dydrogesterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medroxyprogesterone Acetate (Experimental): EH patients will take MPA (Medroxyprogesterone Acetate) 10mg daily from tenth day of menstruation for 15 days for 3months. Endometrial Biopsy (Pipelle) will be performed every 3 months to examine the endometrium. All of the findings will be recorded.
  Interventions: Drug: Medroxyprogesterone Acetate
- dydrogesterone (Experimental): EH patients will take dydrogesterone 10 mg, 2 tablets twice daily from tenth day of menstruation for 15 days for 3-6 months. Endometrial Biopsy (Pipelle) will be performed every 3-month to examine the endometrium. All of the findings will be recorded.
  Interventions: Drug: Dydrogesterone 10 MG

INTERVENTIONS:
Drug: Medroxyprogesterone Acetate — At a dosage of 10mg/day
  Other Names: Provera
  Arms: Medroxyprogesterone Acetate
Drug: Dydrogesterone 10 MG — At a dosage of 20 mg/day
  Other Names: Duphaston
  Arms: dydrogesterone

SUMMARY:
To compare the efficacy of Medroxyprogesterone Acetate with dydrogesterone in patients having endometrial hyperplasia (EH) without atypia.

DETAILED DESCRIPTION:
Patients pathologically diagnosed with nonatypical simple or complex EH will be enrolled. Exclusion criteria include malignancy, liver disease or liver tumor (benign or malignant), kidney disease or kidney tumor (benign or malignant), any contradictions against progesterone, history of endometrial atypical hyperplasia or endometrial cancer, any progesterone-dependent tumors, ask for other treatment.

A detailed history including menstruation, fertility, other diseases and family history will be collected. Basic information including age, waist circumstances, hip circumstances and blood pressure will also be collected. Blood tests including fasting blood glucose (FBG), postprandial blood glucose (PBG), fasting insulin (FINS), SHBG, sex hormone levels, blood lipids, liver and kidney functions will be performed before taking progesterone orally.

All enrolled and consent informed patients will be randomized into two groups, A and B, using computer-generated random numbers. Patients in group A will orally take MPA (Medroxyprogesterone Acetate) (angonghuangtitong, Xianju pharmaceuticals, China)10mg daily from tenth day of menstruation for 15 days for 3-6months. While patients in group B will take dydrogesterone (duphaston; Abbott Healthcare Products B.V, the Netherlands) 10 mg, 2 tablets twice daily from fifth day of menstruation for 20 days for 3-6 months. Endometrial Biopsy (Pipelle) will be performed every 3 months to examine the endometrium.

Complete response (CR) is defined as the reversion of EH to proliferative or secretory endometrium; partial response (PR) is defined as regression to disordered proliferative endometrium (DPE) or simple hyperplasia without atypic (only for complex hyperplasia); no response (NR) is defined as the persistence of the disease; and progressive disease (PD) is defined as the progression of endometrial lesions.

Another 3-month therapy will be continued if the patients get NR. The longest treatment periods will be 6 months. If the patient gets PD or NR after 6 months therapy, new options must be put.

At least 3-month maintenance therapy will be recommended for patients get CR. And all of the enrolled patients will be followed up for 2 years. All data of the therapy, reverse events, side effects, pregnancy and long-term outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of endometrial hyperplasia without atypia;
* Consent informed and signed;
* Able to follow treatment and take therapy in Obstetrics and Gynecology of Fudan University

Exclusion Criteria:

* Liver disease or liver tumor (benign or malignant)
* Kidney disease or kidney tumor (benign or malignant)
* Other malignancies in reproductive organs
* Breast cancer or other progesterone-dependent tumors
* History of endometrial atypical hyperplasia or endometrial cancer
* Any contradictions against progesterone
* Under treatment of progestin therapy or oral conceptive drugs one month before enrollment.
* Pregnancy or suspicion of pregnancy
* Ask for other treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 471 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (CR) rates | From date of randomization until the date of CR, assessed up to 6 months
  The CR rates will be calculated after 3 and 6-month therapy based on the following formula: (Number of participants who got CR)/(All enrolled participants). The CR rates will be compared between two therapies (MPA VS dydrogesterone), also between two lesions (SH VS CH).

SECONDARY OUTCOMES:
Median time of pathological complete response (CR) | From date of randomization until the date of CR, assessed up to 6 months
  Median time of histologic regression from endometrial hyperplasia without atypia to normal endometrium, and comparison will be performed between two treatments and two lesions (SH vs CH).
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 2 years after the treatment for each patient
  Adverse events related with MPA (Medroxyprogesterone acetate
  ) or dydrogesterone include acne, irregular bleeding, breast tenderness, decreased scalp hair, difficulty falling or remaining asleep, stomach pain, and weight loss or gain, depression and mood changes. Severe side effects include thrombus and impaired liver and kidney function. The investigators will record any symptoms, evaluate the correlation and count the events. And comparison will be performed between two treatments and two lesions (SH vs CH).
Relapse rates | up to 2 years after the treatment for each patient
  All enrolled patients will be followed up for 2 years. During the following-up period, if patients recur after complete regression, they will be counted and the number of recurrence will be divided by number of patients followed up, then we can get the relapse rates.Comparison will be performed between two treatments and two lesions (SH vs CH).
Rate of pregnancy | up to 2 years after the treatment for each patient
  For patients have a desire for fertility, pregnancies, births and related outcomes will be counted, and the rate of pregnancy will be counted as number of pregnancies/ number of patients trying to fertility in the following period. Comparison will be performed between two treatments and two lesions (SH vs CH).
Compliance | up to 2 years after the treatment for each patient
  The investigators designed a questionnaire to evaluate the compliance through treatment. Comparison will be performed between two treatments and two lesions (SH vs CH).
cost | From date of randomization until the date of CR, assessed up to 6 months
  Treatment-related cost in each patient during the period beginning from randomization to the date of CR.Comparison will be performed between two treatments and two lesions (SH vs CH).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, PhD, Study Chair — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China